CLINICAL TRIAL: NCT02133378
Title: Prospective, Randomized Clinical Trial of the Hemopatch Topic Hemostatic in Cardiac Surgery.
Brief Title: Prospective Clinical Trial of the Hemopatch Topic Hemostatic in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiochirurgia E.H. (Other)
Responsible Party: Principal Investigator, Luca Weltert, Dr. Luca Weltert, Cardiochirurgia E.H.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-01
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Bleeding
Keywords: Bleeding; Hemostatic
MeSH Terms: conditions — Hemorrhage | interventions — Desiccation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemopatch (Experimental): Use of Hemopatch on bleeding spot
  Interventions: Device: Hemopatch
- Control (Sham Comparator): Traditional techniques hemostasis (dry or wet gauze compression or similar)
  Interventions: Behavioral: Traditional Hemostasis Techniques (dry or wet gauze compression or similar)

INTERVENTIONS:
Device: Hemopatch — Baxter Hemopatch
  Arms: Hemopatch
Behavioral: Traditional Hemostasis Techniques (dry or wet gauze compression or similar)
  Arms: Control

SUMMARY:
A new topical hemostatic agent composed of a specifically-formulated porous collagen matrix, coated on one side with a thin protein bonding layer (known as NHS-PEG) has been reported to be extremely effective, in addition to traditional means, in terminating bleeding during cardiac operations with control rates as high as 97,5%. The investigators compared such hemostatic agent (Hemopatch; Baxter Inc, Deerfield, IL) with traditional optimized hemostasis routine.

Following sample size calculation, in a prospective randomized study design, 100 patients will be treated with Hemopatch and 100 patients will receive traditional optimized hemostasis routine (comparison group).

To make the two cohorts as comparable as possible enrollment will be restricted to moderately bleeding vascular anastomosis of Dacron grafts to ascending aorta or moderately bleeding transversal aortotomy.

Study endpoints are the following: rate of successful intraoperative hemostasis (identified by cessation of bleeding in less than 3 minutes from application) and time required for hemostasis; overall postoperative bleeding; rate of transfusion of blood products; rate of surgical revision for bleeding; postoperative morbidity; and intensive care unit stay.

ELIGIBILITY:
Inclusion Criteria:

* Surgery on Ascending Aorta with Dacron Graft or transverse Aortotomy
* Moderate bleeding

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Successful Hemostasis in under 3 minutes | 3 minutes
  Application of Hemopatch or traditional techniques (compression with dry or wet gauze or similar) are considered successful if hemostasis is reached in under 3 minutes

SECONDARY OUTCOMES:
Post Operative Blood Loss | 6 hours
  Blood loss in the first 7 hours postoperatively

OTHER OUTCOMES:
Allogeneic Blood Transfusion | 4 days
  Allogeneic Blood Transfusion in the first 4 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- European Hospital, Rome, Italy

REFERENCES:
- [Background] Nasso G, Piancone F, Bonifazi R, Romano V, Visicchio G, De Filippo CM, Impiombato B, Fiore F, Bartolomucci F, Alessandrini F, Speziale G. Prospective, randomized clinical trial of the FloSeal matrix sealant in cardiac surgery. Ann Thorac Surg. 2009 Nov;88(5):1520-6. doi: 10.1016/j.athoracsur.2009.07.014. PMID 19853105